CLINICAL TRIAL: NCT03238950
Title: In Cricothyroidotomy Training for Physicians Does Simulated Practice With Tissue Specimens Produce Better Outcomes Than Using Synthetics Manikins?
Brief Title: Cricothyroidotomy Training for Physicians Outcomes Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has never actually started as waiting on funding
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017SUR96
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Porcine Group (Other): Training conducted on Porcine model
  Interventions: Other: Porcine model
- Synthetic (Other): Training conducted on synthetic model
  Interventions: Other: Synthetic model

INTERVENTIONS:
Other: Porcine model — participants to conduct training on porcine model
  Arms: Porcine Group
Other: Synthetic model — participants to conduct training on synthetic model
  Arms: Synthetic

SUMMARY:
This study will assess whether the type of simulation model used in cricothyroidotomy training has an effect on the subsequent confidence and competence in the procedure.

DETAILED DESCRIPTION:
This is a Pilot study - prospective randomised controlled trial involving:

1. Assessment of ability to complete a surgical cricothyroidotomy
2. Completion of questionnaire prior to training and prior to assessment

Prior to beginning training, questionnaires will be completed by all participants asking their level of previous training. Current confidence level for completion of cricothyroidotomy will be marked on a visual analogue scale (VAS).

Training will then be completed with each group using the appropriate manikin type - porcine or synthetic. This will consist of didactic information on the procedure delivered via recorded information to standardise this initial training, and then proceeding to supervised practice of the procedure for two occasions. This will be completed by the same trainer, with the same information given to both groups. Questions to clarify how to perform the procedure will be permitted.

The second questionnaire will be given to the trainees on completion of training to mark on a visual analogue scale their confidence level at this point.

Assessment will then be completed later the day comprising of assessment of completion of surgical cricothyroidotomy using a porcine manikin with skin overlying. This will be different to the porcine manikin used for training. The assessment will time the trainees from start to completion of airway insertion, as well as a checklist of activities to be achieved. The porcine manikins will then be dissected to identify if correct location for insertion was achieved and complications. The same amount of time will be given between groups training and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Medically trained healthcare professionals working in Anaesthetics, Emergency Medicine or General Surgery as these doctors may be expected to complete a surgical cricothyroidotomy despite infrequently performing the procedure.
* The healthcare professionals can be from Foundation Year 1 to before Certificates of Completion of Training (CCT). Those who are out of training and are not yet at consultant level are also eligible.
* Able to provide informed consent.

Exclusion Criteria:

• Healthcare professionals who already complete surgical airways on a regular basis (e.g. Ear Nose Throat or Maxillofacial trainees) as these doctors may already be competent prior to training.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to successfully complete surgical cricothyroidotomy on a prepared porcine specimen. | 1 day
  time

SECONDARY OUTCOMES:
Success rate for cricothyroidotomy | 1 day
  subjective reporting of confidence through questionnaire
Complication rate for cricothyroidotomy | 1 day
  subjective reporting of confidence through questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Helme, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan